CLINICAL TRIAL: NCT05318833
Title: A Phase I Clinical Study on the Safety, Tolerability, Pharmacokinetics and Efficacy of HRS7415 Tablets in Patients With Advanced Malignant Tumors
Brief Title: A Study of HRS7415 Tablets in Patients With Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS7415-I-101
Record Dates: First submitted 2022-03-18; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Advanced Malignant Tumor

STUDY DESIGN:
Intervention Model Description: The study was divided into two phases, the dose escalation phase and the dose extension phase of HRS7415 in subjects with advanced malignant tumors.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS7415 (Experimental)
  Interventions: Drug: HRS7415

INTERVENTIONS:
Drug: HRS7415 — Drug: HRS7415

SUMMARY:
This study is a multicenter, open phase I clinical study of dose escalation and dose extension of HRS7415 in subjects with advanced malignant tumors. To evaluate the safety, tolerability, pharmacokinetics and efficacy of HRS7415 tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects volunteered to participate in the clinical study, understood the study procedure and was able to sign informed consent in person.
2. 18 to 75 years old, male or female.
3. ECOG Performance Status of 0 or 1.
4. The estimated survival time is ≥12 weeks.
5. Subjects with advanced or metastatic malignancy confirmed by histopathology or cytology.
6. Solid tumor subjects had measurable lesions that met RECIST 1.1 criteria.
7. Adequate hematology and terminal organ function, with vital organ function meeting the upper and lower limits required by the protocol.
8. Male subjects and fertile female subjects must agree to use medically approved contraception during the study period and for 6 months following the study; Fertile female subjects must have a negative serum human chorionic gonadotropin (HCG) test within 7 days prior to initial dosing and must be non-lactation blood pregnancy test must be negative and not lactation.

Exclusion Criteria:

1. Subjects plan to receive any other antitumor therapy during the study period.
2. Subjects received chemotherapy, radiotherapy, biotherapy, targeted therapy, or immunotherapy within 4 weeks prior to initial dosing.
3. Major surgery other than diagnosis or biopsy was performed within 4 weeks prior to initial dosing.
4. Received any other investigational drug or treatment that is not on the market within 4 weeks prior to initial dosing.
5. The damage caused by any previous antineoplastic therapy has not recovered to grade ≤1.
6. Imaging diagnosis showed tumor lesion or meningeal metastasis in the brain.
7. Active heart disease in the 6 months prior to initial dosing.
8. Had other malignancies within 5 years prior to first dosing.
9. Subjects with poorly controlled hypertension and a previous history of hypertensive crisis or hypertensive encephalopathy.
10. Having one of several factors affecting oral medication or having active gastrointestinal disease or other medical conditions that may result in significant influence on drug absorption, distribution, metabolism or excretion;
11. Active hepatitis B and C;
12. Serious infections that require intravenous antibiotics, antivirals or antifungals to control;
13. History of immune deficiency or organ transplantation;
14. Comorbidities or any other conditions that, in the investigator's judgment, seriously endanger patient safety or prevent patients from completing the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | From the beginning of first patient in (FPI) to the end of dose escalation phase up to approximately 10 months
maximum tolerated dose (MTD) | From the beginning of first patient in (FPI) to the end of dose escalation phase up to approximately 10 months
Phase II recommended dose (RP2D) | From the beginning of first patient in (FPI) to the end of dose escalation phase up to approximately 10 months

SECONDARY OUTCOMES:
Incidence, severity, duration, and association of adverse events (AE) and severe adverse events (SAE) with the study drug, in addition to abnormalities in vital signs, electrocardiogram, and laboratory tests | From the beginning of first patient in (FPI) to the end of study up to approximately 2 years
Single dose parameters: Peak plasma concentration (Cmax) of HRS7415 and its main metabolite after single dosing | From the beginning of first patient in (FPI) to the end of study up to approximately 2 years
Single dose parameters: Time to peak (Tmax) of HRS7415 and its main metabolite after single dosing | From the beginning of first patient in (FPI) to the end of study up to approximately 2 year
Single dose parameters: Area under the curve from 0 to the last measurable concentration time point t (AUC0-t) of HRS7415 and its main metabolite after single dosing (if applicable) | From the beginning of first patient in (FPI) to the end of study up to approximately 2 years
Single dose parameters: Area under the time curve from 0 to infinity (AUC0-inf) of HRS7415 and its main metabolite after single dosing (if applicable) | From the beginning of first patient in (FPI) to the end of study up to approximately 2 years
Single dose parameters: Half-value period (t1/2) of HRS7415 and its main metabolite after single dosing (if applicable) | From the beginning of first patient in (FPI) to the end of study up to approximately 2 years
Single dose parameters: Apparent volume of distribution (Vz/F) of HRS7415 and its main metabolite after single dosing (if applicable) | From the beginning of first patient in (FPI) to the end of study up to approximately 2 years
Single dose parameters: Apparent clearance (CL/F) of HRS7415 and its main metabolite after single dosing (if applicable) | From the beginning of first patient in (FPI) to the end of study up to approximately 2 years
Multiple dose parameters: Steady state peak concentration (Cmax，ss) of HRS7415 and its main metabolite after multiple dosing | From the beginning of first patient in (FPI) to the end of study up to approximately 2 years
Multiple dose parameters: Time to peak (Tmax, ss) of HRS7415 and its main metabolite after multiple dosing | From the beginning of first patient in (FPI) to the end of study up to approximately 2 years
Multiple dose parameters: Steady valley concentration (Cmin，ss) of HRS7415 and its main metabolite after multiple dosing | From the beginning of first patient in (FPI) to the end of study up to approximately 2 years
Multiple dose parameters: Area under steady-state drug concentration-time curve (AUCss) of HRS7415 and its main metabolite after multiple dosing | From the beginning of first patient in (FPI) to the end of study up to approximately 2 years
Multiple dose parameters: Drug storage ratio (Rac) of HRS7415 and its main metabolite after multiple dosing | From the beginning of first patient in (FPI) to the end of study up to approximately 2 years
Efficacy endpoints: Objective response rate (ORR) | From the beginning of first patient in (FPI) to the end of study up to approximately 2 years
Efficacy endpoints: Disease control rate (DCR) | From the beginning of first patient in (FPI) to the end of study up to approximately 2 years
Efficacy endpoints: Duration of response (DoR) | From the beginning of first patient in (FPI) to the end of study up to approximately 2 years
Efficacy endpoints: Progression-free survival (PFS) | From the beginning of first patient in (FPI) to the end of study up to approximately 2 years

IPD SHARING:
Plan to Share IPD: Undecided